CLINICAL TRIAL: NCT01163097
Title: An Open-label, Randomized, Parallel-Design Study to Characterize the Effect of Heparin on Palifermin Activity in Healthy Adult Subjects
Brief Title: Study to Characterize the Effect of Heparin on Palifermin Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070278
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Fibroblast Growth Factor 7; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Palifermin 40 µg/kg and heparin IV infusion (Experimental): Treatment A: palifermin 40 µg/kg/day for three consecutive days as IV bolus injections and continuous heparin IV infusion
  Interventions: Drug: Palifermin; Drug: Heparin
- Palifermin 40 µg/kg (Experimental): Treatment B: palifermin 40 µg/kg/day for three consecutive days as IV bolus injections
  Interventions: Drug: Palifermin
- Control group without any treatment (No Intervention): Treatment C: control group without any treatment administered.

INTERVENTIONS:
Drug: Palifermin — 40 µg/kg IV bolus injections for three consecutive days
  Arms: Palifermin 40 µg/kg; Palifermin 40 µg/kg and heparin IV infusion
Drug: Heparin — Heparin continuous IV infusion
  Arms: Palifermin 40 µg/kg and heparin IV infusion

SUMMARY:
The purpose of this study is to evaluate the effect of a continuous intravenous infusion of unfractionated heparin on the multiple-dose pharmacodynamics of palifermin in healthy adult subjects.

DETAILED DESCRIPTION:
The planned study is designed to characterize the impact of heparin on the biologic activity of palifermin and assess the impact of the combination of palifermin and heparin on tolerability. Approximately forty-three (43) eligible healthy adult men and oophorectomized or postmenopausal women between 18-45 years of age will be assigned to one of three treatment groups where treatment group A will receive a daily dose of palifermin 40 µg/kg for three consecutive days as intravenous (IV) bolus injections and continuous heparin IV infusion, treatment B will receive a daily dose of palifermin 40 µg/kg for three consecutive days as IV bolus injections and treatment C will be a control group without any treatment administered. The subjects will be randomized in a 20:15:8 ratio (Treatment A:B:C).

The study consists of a up to 21-days screening period, a 5-days treatment period and a up to 45-days follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or postmenopausal or oophorectomized women.
* Subjects should have a Body Mass Index between 19 and 30 inclusive.
* A negative screen for drug abuse, tobacco use and alcohol breath test.
* Subjects should be willing to be resident in the research facility for up to 6 nights and return to the research facility for scheduled study and follow-up procedures.
* Men must agree for the duration of the study to use an appropriate method of birth control

Exclusion Criteria:

* History or evidence of clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* History or evidence of any oral mucosal disease that may affect mucosal keratinocyte proliferation.
* Evidence or history of thrombocytopenia, heparin-induced thrombocytopenia or other contraindications to heparin (e.g. recent surgeries).
* Known hypersensitivity to heparin or topical or injectable local anesthetic.
* Known allergies to Escherichia coli-derived products or allergies to palifermin or its excipients.
* Use of medications (except vitamins, hormonal replacement therapy and topical medications) within 10 days of admission to research facility.
* Blood donation within 8 weeks prior to dosing of investigational drug.
* History of hypertension, clinically significant bleeding, gastrointestinal ulcers, arteriovenous malformation (AVM), aneurysm, or other vascular malformation.
* History of coagulopathy, bleeding disorders or abnormal platelet counts.
* History of malignancy of any type, other than surgically excised non-melanoma skin cancers or in situ cervical cancer.
* For males, past history of epididymitis.
* Known alcohol abuse or use of illicit drugs within 12 months prior to admission to the research facility.
* History of smoking or using smokeless tobacco within the past year before admission to the research facility.
* Any other condition that might reduce the chance of obtaining data (eg, known poor compliance) required by the protocol or that might compromise the ability to give informed consent.
* Previous participation in a palifermin study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten de Chateau, MD PhD, Study Director — Swedish Orphan Biovitrum
Locations (1):
- New Orleans Center for Clinical Research (NOCCR), Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Yang BB, Gillespie B, Smith B, Smith W, Lissmats A, Rudebeck M, Kullenberg T, Olsson B. Pharmacokinetic and pharmacodynamic interactions between palifermin and heparin. J Clin Pharmacol. 2015 Oct;55(10):1109-18. doi: 10.1002/jcph.516. Epub 2015 May 28. PMID 25880826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, randomized, parallel-design, Phase I study in healthy adult subjects was performed in 1 center (New Orleans Center for Clinical Research, Knoxville, TN, USA) between July and December 2010.
Pre-assignment Details: Subjects randomized to receive palifermin in combination with heparin did first enter a titration period where they received titrated heparin doses to achieve an aPTT of 1.5 to 2.0 × baseline. Subjects who could not be successfully titrated within the heparin titration period were discontinued, and did not enter the palifermin treatment period.
Groups:
- Palifermin - Heparin: Treatment A: palifermin 40 µg/kg/day for three consecutive days as IV bolus injections and continuous heparin IV infusion
- Palifermin Alone: Treatment B: palifermin 40 µg/kg/day for three consecutive days as IV bolus injections
- Untreated Control: Treatment C: control group without any treatment administered
Period: Overall Study
Arm/Group | Palifermin - Heparin | Palifermin Alone | Untreated Control
Started | 20 (15 subjects were successfully titrated and entered the palifermin treatment) | 16 | 8
Completed | 14 | 16 | 8
Not Completed | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palifermin - Heparin | Palifermin Alone | Untreated Control | Total
Number analyzed (Participants) | 15 | 16 | 8 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 8 | 39
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (5.29) | 32.9 (7.82) | 22.8 (3.62) | 28.1 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 15 | 16 | 8 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 16 | 8 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 12 | 14 | 7 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 8 | 39
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 24.95 (2.144) | 26.08 (2.111) | 25.98 (3.185) | 25.62 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Ratio to Baseline of Epithelial Cell Proliferation as Assessed by Ki67 Staining of Buccal Mucosal Tissue.
Description: This outcome is a measure of the palifermin effect on the buccal mucosal cells. Ki67 is a measure of proliferation of cells in the buccal mucosa. This measure assess the number of cells per millimeter (mm) before and after palifermin treatment.
Time Frame: Day 4
Population: The pharmacodynamic population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B), or who had a set zero point (Treatment C) and had both baseline and Day 4 buccal biopsy samples collected. This analysis was only performed for Treatment A relative to Treatment B as per study plan.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 14 | 16
ratio | 0.267 [0.173 to 0.361] | 0.414 [0.326 to 0.502]
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; H0: mean ratio<0.7 or mean ratio>1.43; H1: 0.7< mean ratio <1.43 Sample size calculation assumed change in Ki67 expression following palifermin administration would not be affected by co-administration of heparin. With n=26 (13 + 13), an approx. 80% probability that the 90% CI of the ratio of geometric means of Ki67 for palifermin when co-administered with heparin compared to palifermin alone would fall in the interval (0.7, 1.43). This assumed a Coefficient of Variation (CV) for Ki67 of 31%; Test type: Non-Inferiority or Equivalence — The equivalence of the treatments was assessed using the 90% confidence interval (CI) of the geometric mean ratio for Ki67. The lower bound of the CI needed to be greater than 0.70 and the upper bound needed to be below 1.43 for the treatments to be considered equivalent; ANCOVA; ANCOVA was used to estimate the treatment effect and the Schuirmann's two one-sided test was used to test for statistical equivalence; Geometric mean ratio = 0.863, 90% CI 2-sided [0.759 to 0.982]

2. Primary Outcome: Incidence of Grade 2 or Higher Specific Skin-related Adverse Events.
Description: Incidence of grade 2 or higher specific skin-related treatment emergent adverse events following palifermin administration was calculated for subjects in treatment groups A and B. Incidence was calculated by treatment as number of subjects with grade 2 or higher specific skin-related AEs divided by the total number of subjects.
  The Common Terminology Criteria for Adverse Events (CTCAE v3.0) for Dermatology/Skin was used to determine the toxicity grade for a skin-related adverse event. (http://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/ctcaev3.pdf)
Time Frame: Day 45
Population: The safety population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B), or who had a set zero point (Treatment C). This outcome was assessed for Treatment A and B only as per study plan.
Measure: Number; unit: proportion of participants
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
proportion of participants | 0 | 0.0625

3. Primary Outcome: Ratio to Baseline of Amylase
Description: Ratio to baseline amylase at Day 5 was calculated as Day 5 amylase divided by baseline amylase.
Time Frame: Day 5
Population: The safety population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B) or who had a set zero point (Treatment C). This outcome was assessed for Treatment A and B only as per study plan.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
ratio | 0.242 [0.111 to 0.372] | 0.547 [0.420 to 0.673]
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; 80% power achieved for detecting a 20% increase (or 17% reduction) when Treatment A was compared to Treatment B; assuming that the coefficient of variation of amylase would be 14% (as observed in other study); Test type: Superiority or Other; ANCOVA; ANCOVA (with dependent variable:natural log of the ratio to baseline, independent variable:treatment, covariate:natural log of the baseline value); Geometric mean = 0.737, 95% CI 2-sided [0.614 to 0.885]

4. Primary Outcome: Ratio to Baseline of Lipase.
Description: Ratio to baseline lipase at Day 5 was calculated as Day 5 lipase divided by baseline lipase.
Time Frame: Day 5
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
ratio | -0.487 [-0.873 to -0.100] | 0.499 [0.125 to 0.873]
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; 80% power achieved for detecting a 70% increase (or 41% reduction) when Treatment A was compared to Treatment B; assuming that the coefficient of variation of lipase would be 49% (as observed in other study); Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Geometric mean = 0.373, 95% CI 2-sided [0.216 to 0.645]

5. Primary Outcome: Ratio to Baseline of Protein/Creatinine
Description: Protein/creatinine ratio is the urinary protein (mg) divided by the urinary creatinine (g) result.
  Ratio to baseline protein/creatinine ratio was calculated as protein/creatinine ratio at specified day divided by baseline protein/creatinine ratio.
Time Frame: Day 4
Population: The safety population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B) or who had a set zero point (Treatment C). This outcome was assessed for Treatment B and C only as per study plan.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 0.076 [-0.058 to 0.211] | 0.104 [-0.087 to 0.296]
Statistical Analysis 1: Comparison: Palifermin Alone vs Untreated Control; 80% power achieved for detecting a 140% increase with 13 and 6 subjects (respectively) when Treatment B was compared to Treatment C; assuming that the coefficient of variation of the protein/creatinine ratio would be 67% (Ginsberg et al 1983); Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Geometric mean = 0.972, 95% CI 2-sided [0.768 to 1.231]

6. Secondary Outcome: Palifermin Pharmacokinetic (PK) Parameters: Clearance (CL)
Description: Blood samples for palifermin PK was collected pre-dose on Days 1 and 3 of the treatment period; 2, 5, 15 and 30 minutes; and 1, 2, 4, 6, 12, 18 and 24 hours after the Day 1 and Day 3 dose of palifermin.
  Descriptive PK parameters for palifermin CL for subjects assigned to Treatment A and Treatment B was determined by linear/log trapezoidal method. Parameters was calculated from individual subject serum concentration-time data using actual subject blood collection times. Serum concentrations reported below the lower limit of quantification (LLOQ) was treated as zero.
Time Frame: Day 1
Population: The pharmacokinetics (PK) population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B) and at least one post dose PK serum sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mL/hr/kg)
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
(mL/hr/kg) | 121.1 (29.1) | 527.8 (33.5)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p < 0.0001, ANOVA

7. Secondary Outcome: Palifermin PK Parameters: CL
Description: as for outcome 6
Time Frame: Day 3
Population: The pharmacokinetics population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B) and at least one post dose PK serum sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mL/hr/kg)
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
(mL/hr/kg) | 121.9 (20.4) | 524.3 (59.4)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p < 0.0001, ANOVA

8. Secondary Outcome: Palifermin PK Parameters: Area Under the Serum Curve (AUC) (0-24)
Description: Blood samples for palifermin PK was collected pre-dose on Days 1 and 3 of the treatment period; 2, 5, 15 and 30 minutes; and 1, 2, 4, 6, 12, 18 and 24 hours after the Day 1 and Day 3 dose of palifermin.
  Descriptive pharmacokinetic parameters for palifermin AUC(0-24) was determined by linear/log trapezoidal method. Parameters was calculated from individual subject serum concentration-time data using actual subject blood collection times. Serum concentrations reported below the lower limit of quantification (LLOQ) was deleted from calculation.
Time Frame: Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
ng*hr/mL | 330.1 (26.9) | 75.80 (37.1)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p < 0.0001, ANOVA

9. Secondary Outcome: Palifermin PK Parameters: AUC (0-24)
Description: as for outcome 8
Time Frame: Day 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
ng*hr/mL | 328.1 (20.4) | 76.26 (36.3)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p < 0.0001, ANOVA

10. Secondary Outcome: Palifermin PK Parameters: Estimated Concentration at Time 0 (C0)
Description: Blood samples for palifermin PK was collected pre-dose on Days 1 and 3 of the treatment period; 2, 5, 15 and 30 minutes; and 1, 2, 4, 6, 12, 18 and 24 hours after the Day 1 and Day 3 dose of palifermin.
  Descriptive pharmacokinetic parameters for palifermin C0 was determined by linear/log trapezoidal method. Parameters was calculated from individual subject serum concentration-time data using actual subject blood collection times. Serum concentrations reported below the lower limit of quantification (LLOQ) was treated as zero.
Time Frame: Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
ng/mL | 229.1 (116.6) | 584.7 (111.9)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p = 0.4123, ANOVA

11. Secondary Outcome: Palifermin PK Parameters: C0
Description: as for outcome 10
Time Frame: Day 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
ng/mL | 361.0 (92.3) | 563.2 (105.7)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p = 0.9944, ANOVA

12. Secondary Outcome: Palifermin PK Parameters: Apparent Volume of Distribution at Steady State (Vss)
Description: Blood samples for palifermin PK was collected pre-dose on Days 1 and 3 of the treatment period; 2, 5, 15 and 30 minutes; and 1, 2, 4, 6, 12, 18 and 24 hours after the Day 1 and Day 3 dose of palifermin (Treatment A and Treatment B only).
  Descriptive pharmacokinetic parameters for palifermin Vss was determined by linear/log trapezoidal method. Parameters was calculated from individual subject serum concentration-time data using actual subject blood collection times. Serum concentrations reported below the lower limit of quantification (LLOQ) was treated as zero.
Time Frame: Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
mL/kg | 411.5 (42.4) | 1586 (48.1)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p < 0.0001, ANOVA

13. Secondary Outcome: Palifermin PK Parameters: Vss
Description: as for outcome 12
Time Frame: Day 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/Kg
Arm/Group | Palifermin - Heparin | Palifermin Alone
Number analyzed (Participants) | 15 | 16
mL/Kg | 361.7 (28.0) | 1318 (64.4)
Statistical Analysis 1: Comparison: Palifermin - Heparin vs Palifermin Alone; Test type: Superiority or Other; p < 0.0001, ANOVA

14. Secondary Outcome: Subject Incidence of Treatment-emergent Adverse Event
Description: Adverse events (AE) was considered treatment emergent if the AE started after the time of heparin titration (Treatment A), palifermin dosing on Day 1 (Treatment B), or set zero point (Treatment C).
Time Frame: Day 45
Population: The safety population consist of all randomized subjects who received at least one dose of palifermin (Treatment A or B) or who had a set zero point (Treatment C)
Measure: Number; unit: participants
Arm/Group | Palifermin - Heparin | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 14 | 16 | 8
participants | 9 | 8 | 3

15. Secondary Outcome: Subject Incidence of Proteinuria
Description: Protein/creatinine ratio is the urinary protein (mg) divided by the urinary creatinine (g) result at the specified time point.
  Incidence of proteinuria defined as urinary protein/creatinine ratio exceeding 200 mg/g was calculated at Day 4 and overall at any time point. Incidence was calculated by treatment as number of subjects with proteinuria divided by the total number of subjects.
Time Frame: Day 4
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
participants | 0 | 0

16. Secondary Outcome: Ratio to Baseline of Protein/Creatinine
Description: as for outcome 5
Time Frame: Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.00 (0.00) | 1.00 (0.00)

17. Secondary Outcome: Ratio to Baseline of Protein/Creatinine
Description: as for outcome 5
Time Frame: Day 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.0 (0.42) | 1.0 (0.13)

18. Secondary Outcome: Ratio to Baseline of Protein/Creatinine
Description: as for outcome 5
Time Frame: Day 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.1 (0.51) | 1.1 (0.33)

19. Secondary Outcome: Ratio to Baseline of Albumin/Creatinine
Description: The albumin/creatinine ratio is the urinary albumin (mg) divided by the urinary creatinine (g) result at the specified time point.
  Ratio to baseline was calculated as albumin/creatinine ratio at specified day divided by baseline albumin/creatinine ratio.
Time Frame: Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.00 (0.000) | 1.00 (0.000)

20. Secondary Outcome: Ratio to Baseline of Albumin/Creatinine
Description: as for outcome 19
Time Frame: Day 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.05 (0.373) | 0.95 (0.230)

21. Secondary Outcome: Ratio to Baseline of Albumin/Creatinine
Description: as for outcome 19
Time Frame: Day 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.16 (0.391) | 0.99 (0.268)

22. Secondary Outcome: Ratio to Baseline of Albumin/Creatinine
Description: as for outcome 19
Time Frame: Day 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Palifermin Alone | Untreated Control
Number analyzed (Participants) | 16 | 8
ratio | 1.56 (1.610) | 1.25 (0.484)

ADVERSE EVENTS:
Time Frame: From signing of informed consent to subject´s end of study.
Arm/Group | Palifermin - Heparin | Palifermin Alone | Untreated Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 9/20 | 9/16 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palifermin - Heparin (N=20) | Palifermin Alone (N=16) | Untreated Control (N=8)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 6 (8) | 3 (5)
Headache (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 3 (3) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Poor venous access (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 90 days). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.